CLINICAL TRIAL: NCT03945994
Title: Connecting People Implementation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of York (Other)
Responsible Party: Principal Investigator, Martin Webber, PhD, Professor of Social Work, Department of Social Policy & Social Work, University of York
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 225304
Record Dates: First submitted 2018-05-01; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Social Isolation; Mental Health Wellness 1; Social Interaction
Keywords: Improve Social Capital; Improve mental health
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: This study will use multiple methods to answer our research questions. It will consist of:
  1. a natural experiment in the form of a non-randomised wait-list controlled pre-post study to evaluate the outcomes of the CP programme, when implemented in CMHTs, in contrast to standard care; and
  2. an evaluation of the implementation tools using a standardised tool and qualitative approaches to understand the barriers and facilitators of implementation in the different sites.
Who Masked: Participant, Care Provider
Masking Description: The control group will continue to receive their standard care. A natural experiment in the form of a non-randomised wait-list controlled pre-post study to evaluate the outcomes of the CP programme, when implemented in CMHTs, in contrast to standard care; and
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connecting People Control Group (No Intervention): CMHTs (Community Mental Health Teams) will continue to support people with mental health problems using their standard care.
- Connecting People Intervention Group (Experimental): CMHTs will receive training on how to implement Connecting People programme. They will receive implementation toolkit to improve their practice in contrast to standard care.
  Interventions: Other: Connecting People Intervention

INTERVENTIONS:
Other: Connecting People Intervention — Improve the resourcefulness of social networks of people with mental health problems
  Arms: Connecting People Intervention Group

SUMMARY:
This study aims to investigate if the Connecting People (CP) Programme can be implemented by social care practitioners with high fidelity in community mental health teams (CMHTs) and improve the resourcefulness of social networks of people with mental health problems.

DETAILED DESCRIPTION:
People with mental health problems require a range of support to help them in their recovery. Alongside medical and psychological support, people may need support with engaging in meaningful activities and developing relationships. The focus of this study is on advancing understanding of how services can improve the support they offer to people around social relationships.

In a previous study, a Connecting People programme was developed which supported people to make plans for developing their network of contacts in the community. When delivered fully, it helped people feel more included in society and better able to access advice, information and practical support from people they know.

This research project aims to look at how Connecting People can be effectively established within community mental health teams by social workers trained as part of the 'Think Ahead' initiative. The investigators want to know how to implement the Connecting People programme well, assessing whether tools such as manuals, guidance and specific training help or hinder this process. The investigators want to know when implemented, compared to standard care, whether the programme benefits mental health service users and is cost-effective.

The study will last 15 months and is organised into two phrases:

1. Implementation of the programme in community mental health teams in five areas in England. Outcome data will be collected from each participating team and results will be compared between teams who implemented the programme and those that only offered standard care.
2. Exploration of how successful implementation was across the five areas, using a check-list and in-depth individual and group interviews to understand the features that supported or hindered the process.

ELIGIBILITY:
Inclusion Criteria:

* Adults with mental health problems under CMHTs

Exclusion Criteria:

* Children
* Adults with mental health problems who are not under CMHTs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-07-29 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Resource Generator-UK (RG-UK) | 6 months
  Questionnaire; Measure of access to social capital (knowing people with particular skills or resources within your social network). The name of the scale is the Resource Generator-UK. Example questions include: Do you currently have access to someone who is able to lend you a small amount of money? Do you currently have access to someone who works for the local authority? Answers are 'Yes' or 'No'; though further information is obtained on the relation of the person to the individual. Scale has 27 items and is scored 0-27 with high scores indicating high access to social capital.

SECONDARY OUTCOMES:
Goal Attainment Scaling (GAS) | 6 months
  Questionnaire; GAS is a method of scoring the extent to which service users' individual goals are achieved in the course of intervention. In effect, each service user has their own outcome measure but this is scored in a standardised way as to allow statistical analysis. The name of the scale is the Goal Attainment Scaling (GAS). Importance from 0 (not at all) to 3 (very important). Difficulty: from 0 (not at all) to 3 (very difficult).
Questionnaire about the process of recovery (QPR) | 6 months
  Questionnaire; Measurement of people's perception of their recovery from mental health problems. Items include, for example, 'I feel better abut myself', 'I feel that my life has a purpose'. The scale has 15 items which are answered using a 5-point likert scale from 'strongly disagree' to 'strongly agree'. Responses are scored 1-5 and summed, with totals from 15-75. Higher values represent a better recovery.
EQ-5D-5L | 6 months
  Questionnaire measurement of health related quality of life. The first part comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems and the participant is asked to select the most appropriate for them. The digits for the five dimensions are combined into a 5-digit number that describes the participant's health state. High numbers indicate poor health-related quality of life.
  The second part records the participant's self-rated health on a vertical visual analogue scale (VAS), where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the participant's own judgement from 0-100. High scores indicate better self-rated health.
The Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | 6 months
  Questionnaire measurement of mental well-being. The scale includes 14 items such as 'I've been feeling optimistic about the future'. 'I've been feeling relaxed', 'I've been feeling confident'. Each item is answered using a 5-point likert scale from 'none of the time' to 'all of the time', with values of 1-5 ascribed to each response. The scale is a sum of item values ranging from 15 to 70 with higher values indicating higher mental well-being

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Barber, PhD, Study Director — University of York
Locations (1):
- Tees, Esk And Wear Valley NHS Foundation Trust, Durham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Webber M, Reidy H, Ansari D, Stevens M, Morris D. Enhancing social networks: a qualitative study of health and social care practice in UK mental health services. Health Soc Care Community. 2015 Mar;23(2):180-9. doi: 10.1111/hsc.12135. Epub 2014 Dec 1. PMID 25441461
- [Background] Webber M, Fendt-Newlin M. A review of social participation interventions for people with mental health problems. Soc Psychiatry Psychiatr Epidemiol. 2017 Apr;52(4):369-380. doi: 10.1007/s00127-017-1372-2. Epub 2017 Mar 12. PMID 28286914